CLINICAL TRIAL: NCT05791175
Title: Stress and Tooth Structure Loss in Dental Students. A Prospective, Longitudinal Pilot - Observational Study.
Brief Title: Stress and Tooth Structure Loss in Dental Students.
Acronym: STSLDS
Status: Not yet recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: DresdenStressDentalStudents
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Tooth Wear
MeSH Terms: conditions — Tooth Wear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Teeth scan with intraoral scanner (Trios, 3 Shape, Denmark) — Intraoral scanner will be use to monitor the changes of the teeth over time. Intraoral scanners are devices that capture three-dimensional images of teeth and are used as an alternative to conventional dental impressions.

SUMMARY:
The study is designed as a pilot study. The primary objective of the current study is to collect data on the expression and progression of tooth structure loss in dental students under stressful conditions and different dietary habits using intraoral scanners (IOS). Stress levels will be evaluated using Percived Stress Scale (PSS-10). Eating habits will be queried using reflux and dietary questionnaires. The data obtained will later be used in the case-control design of a multicenter study on the same topic. Conducting the pilot study will allow for a critical evaluation of the study's design, participant retention rate, and recruitment process.

DETAILED DESCRIPTION:
The first scan (baseline: T0) is performed during the Dental Prosthetics I course, at the beginning of the 8th semester. Follow-up scans T1 and T2 are performed at the beginning of the 10th semester and after completion of the state examination. The scans are performed by a study doctor or doctoral student using a digital intraoral scanner (Trios, 3 Shape, Denmark). Accompanying the scanning process, study participants will be asked to complete a questionnaire regarding stress levels (PSS) and dietary habits. A medical history and dental findings are also collected. Each scan will take no longer than 10 minutes. The entire examination will take no longer than 45 minutes. The T0 and T1, T2 scans will be overlaid with evaluation software and compared in terms of tooth wear.

ELIGIBILITY:
Inclusion Criteria:

* At the time of the baseline examination of the study the participants must be dental students and participate in the Dental Prosthetics Course I in the summer semester 2023, at the Dental School of Medical Faculty Carl Gustav Carus at the Technical University of Dresden
* Presence of study teeth (at least one antagonist pair of first molars (16/46 or 26/36).
* Complete dentition, if necessary, dentition with complete gap closure up to the first molar in the maxilla and mandible
* Presence of a canine guidence
* Written informed consent of the participating persons

Exclusion Criteria:

* Age <18 and >40
* Study teeth restored with dentures
* Extensive restorations over 1/3 of the occlusal surface on the study teeth
* Removable dentures
* Ongoing orthodontic treatment
* Existing pregnancy/lactation
* Addiction or other medical conditions that do not allow the subject to understand the nature and scope and possible consequences of the clinical study
* Indications that the participant is unlikely to comply with the protocol.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study participants will be dental students enrolled in Dental Prosthetics Course I at the beginning of the observation period.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-03-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of tooth structure loss and its' progression under stressfull conditons and diverse dietary habits. | 2 years
  Tooth wear will be mesaured in micrometers (µm).

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Passia, Prof. Dr., Study Director — Department of Dental Prosthetics, University Hospital at the Technische Universität Dresden
Locations (1):
- Department of Dental Prosthetics, Dental Division of the University Hospital Carl Gustav Carus at the Technische Universität Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abbasi SZ, Mubeen N, Ayub T, Khan MA, Abbasi Z, Baig N. Comparison of stress levels among medical and dental students in the clinical years of training and their coping strategies. J Pak Med Assoc. 2020 Jun;70(6):1006-1008. doi: 10.5455/JPMA.294959. PMID 32810097
- [Background] Al-Khalifa KS. The Prevalence of Tooth Wear in an Adult Population from the Eastern Province of Saudi Arabia. Clin Cosmet Investig Dent. 2020 Nov 17;12:525-531. doi: 10.2147/CCIDE.S286500. eCollection 2020. PMID 33235511
- [Background] Bartlett D, Ganss C, Lussi A. Basic Erosive Wear Examination (BEWE): a new scoring system for scientific and clinical needs. Clin Oral Investig. 2008 Mar;12 Suppl 1(Suppl 1):S65-8. doi: 10.1007/s00784-007-0181-5. Epub 2008 Jan 29. PMID 18228057
- [Background] Bartlett DW, Coward PY, Nikkah C, Wilson RF. The prevalence of tooth wear in a cluster sample of adolescent schoolchildren and its relationship with potential explanatory factors. Br Dent J. 1998 Feb 14;184(3):125-9. doi: 10.1038/sj.bdj.4809560. PMID 9524373
- [Background] Elani HW, Allison PJ, Kumar RA, Mancini L, Lambrou A, Bedos C. A systematic review of stress in dental students. J Dent Educ. 2014 Feb;78(2):226-42. PMID 24489030
- [Background] Kuhn M, Turp JC. Risk factors for bruxism. Swiss Dent J. 2018 Feb 12;128(2):118-124. doi: 10.61872/sdj-2018-02-369. PMID 29533049
- [Background] Mangano F, Gandolfi A, Luongo G, Logozzo S. Intraoral scanners in dentistry: a review of the current literature. BMC Oral Health. 2017 Dec 12;17(1):149. doi: 10.1186/s12903-017-0442-x. PMID 29233132
- [Background] Marro ML, Aranguiz V, Ramirez V, Lussi A. Prevalence of erosive tooth wear in Chilean adults, 2016: A cross-sectional study. J Oral Rehabil. 2020 Apr;47(4):467-472. doi: 10.1111/joor.12922. Epub 2019 Dec 25. PMID 31834944
- [Background] Mekhemar M, Attia S, Dorfer C, Conrad J. Dental Students in Germany throughout the COVID-19 Pandemic: A Psychological Assessment and Cross-Sectional Survey. Biology (Basel). 2021 Jul 1;10(7):611. doi: 10.3390/biology10070611. PMID 34356466
- [Background] Milosevic A. The problem with an epidemiological index for dental erosion. Br Dent J. 2011 Sep 9;211(5):201-3. doi: 10.1038/sj.bdj.2011.722. PMID 21904350
- [Background] Milosevic Markovic M, Latas MB, Milovanovic S, Poznanovic ST, Lazarevic MM, Karisik MJ, Dordevic J, Mandinic Z, Jovanovic S. Mental Health and Quality of Life among Dental Students during COVID-19 Pandemic: A Cross-Sectional Study. Int J Environ Res Public Health. 2022 Oct 28;19(21):14061. doi: 10.3390/ijerph192114061. PMID 36360939
- [Background] Picos A, Badea ME, Dumitrascu DL. Dental erosion in gastro-esophageal reflux disease. A systematic review. Clujul Med. 2018 Oct;91(4):387-390. doi: 10.15386/cjmed-1017. Epub 2018 Oct 30. PMID 30564013
- [Background] Polmann H, Reus JC, Massignan C, Serra-Negra JM, Dick BD, Flores-Mir C, Lavigne GJ, De Luca Canto G. Association between sleep bruxism and stress symptoms in adults: A systematic review and meta-analysis. J Oral Rehabil. 2021 May;48(5):621-631. doi: 10.1111/joor.13142. Epub 2021 Jan 28. PMID 33377534
- [Background] Schlenz MA, Schlenz MB, Wostmann B, Jungert A, Ganss C. Intraoral scanner-based monitoring of tooth wear in young adults: 12-month results. Clin Oral Investig. 2022 Feb;26(2):1869-1878. doi: 10.1007/s00784-021-04162-6. Epub 2021 Sep 8. PMID 34498100
- [Background] Shellis RP, Addy M. The interactions between attrition, abrasion and erosion in tooth wear. Monogr Oral Sci. 2014;25:32-45. doi: 10.1159/000359936. Epub 2014 Jun 26. PMID 24993256
- [Background] Smith BG, Knight JK. An index for measuring the wear of teeth. Br Dent J. 1984 Jun 23;156(12):435-8. doi: 10.1038/sj.bdj.4805394. No abstract available. PMID 6590081
- [Background] Son K, Lee WS, Lee KB. Effect of Different Software Programs on the Accuracy of Dental Scanner Using Three-Dimensional Analysis. Int J Environ Res Public Health. 2021 Aug 10;18(16):8449. doi: 10.3390/ijerph18168449. PMID 34444195
- [Background] Travassos da Rosa Moreira Bastos R, Teixeira da Silva P, Normando D. Reliability of qualitative occlusal tooth wear evaluation using an intraoral scanner: A pilot study. PLoS One. 2021 Mar 25;16(3):e0249119. doi: 10.1371/journal.pone.0249119. eCollection 2021. PMID 33765042
- [Background] Wetselaar P, Lobbezoo F. The tooth wear evaluation system: a modular clinical guideline for the diagnosis and management planning of worn dentitions. J Oral Rehabil. 2016 Jan;43(1):69-80. doi: 10.1111/joor.12340. Epub 2015 Sep 1. PMID 26333037
- [Background] Wetselaar P, Manfredini D, Ahlberg J, Johansson A, Aarab G, Papagianni CE, Reyes Sevilla M, Koutris M, Lobbezoo F. Associations between tooth wear and dental sleep disorders: A narrative overview. J Oral Rehabil. 2019 Aug;46(8):765-775. doi: 10.1111/joor.12807. Epub 2019 May 12. PMID 31038764
- [Background] Wetselaar P, Wetselaar-Glas MJM, Katzer LD, Ahlers MO. Diagnosing tooth wear, a new taxonomy based on the revised version of the Tooth Wear Evaluation System (TWES 2.0). J Oral Rehabil. 2020 Jun;47(6):703-712. doi: 10.1111/joor.12972. Epub 2020 May 14. PMID 32274827
- [Background] Yu T, Tao DY, Lu HX, Zhu JL, Xie CY, Bartlett D, Feng XP. Prevalence and Associated Factors of Tooth Wear in Shanghai. Chin J Dent Res. 2021 Jun 23;24(2):95-103. doi: 10.3290/j.cjdr.b1530421. PMID 34219442